CLINICAL TRIAL: NCT04189172
Title: Multicenter, International, Prospective, Observational, Study Using Neuro-Patch® in Duraplasty in Neurosurgery (MiDura)
Brief Title: MiDura-Study (Neuro-Patch in Duraplasty)
Acronym: MiDura
Status: Active, not recruiting | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1630
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Meningioma; Tumor, Brain; Chiari Malformation; Vascular Malformation; Hydrocephalus; Tethered Cord; Dural Fistula; Craniotomy; Spinal Surgery; Duraplasty
Keywords: duraplasty; dural substitute; synthetic graft; Neuro-Patch®
MeSH Terms: conditions — Meningioma; Brain Neoplasms; Arnold-Chiari Malformation; Vascular Malformations; Hydrocephalus; Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neuro-Patch: Patients receiving Neuro-Patch® for duraplasty

SUMMARY:
The aim of this study is to collect systematically and proactively data regarding the performance of Neuro-Patch, like complications and handling, under daily clinical practice when used as intended by the manufacturer

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age > 18 years
* Duraplasty using Neuro-Patch® according to the Instructions for Use

Exclusion Criteria:

* Use in infected regions
* Use in open cerebrocranial traumata
* Use in open spina bifida
* Known hypersensitivity to implant materials
* Pregnancy
* Representation by a legal guardian or under involuntary commitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 328 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of complications | until follow-up (up to one year after surgery)
  Incidence of complications, with (potential) causal relationship to Neuro-Patch

SECONDARY OUTCOMES:
Handling measures | Intraoperative
  Evaluation of handling characteristics using a questionnaire containing 5-level Likert scales (excellent, very good, good, fair, poor)
Incidence of complications not related to Neuro Patch | until follow-up (up to one year after surgery)
  Incidence of complications, without causal relationship to Neuro-Patch

CONTACTS AND LOCATIONS:
Locations (4):
- France (2):
  - Service de Neurochirurgie, Hôpital de la Cavale Blanche, Brest
  - Hopital Pierre Wertheimer - HCL, Bron
- Germany (2):
  - Klinik für Neurochirurgie, Universitätsklinikum des Saarlandes, Homburg/Saar
  - Krankenhaus Ludmillenstift, Meppen